CLINICAL TRIAL: NCT00834366
Title: A Study to Compare the Relative Bioavailability of Two 200 Mg Tramadol Hydrochloride Tablet Products Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sybil Robertson, Vice President, Regulatory Affairs, Labopharm Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MDT1-013
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-06-08 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Tramadol

ARMS (2):
- Tramadol HCl 200 mg Film-coated Tablets (Experimental): Single oral administration in fasting conditions of 1x200mg Tramadol HCl 200 mg Film-coated Tablet based on randomization schedule.
  Interventions: Drug: Tramadol HCl
- Tramadol HCl 200 mg Uncoated Tablets (Experimental): Single oral administration in fasting conditions of 1x200mg Tramadol HCl 200 mg Uncoated Tablet based on randomization schedule.
  Interventions: Drug: Tramadol HCl

INTERVENTIONS:
Drug: Tramadol HCl — Single oral administration in fasting conditions of 1x200mg Tramadol HCl 200 mg Film-coated Tablet or Tramadol HCl 200 mg Uncoated Tablets based on randomization schedule.

SUMMARY:
To determine whether the test product, Labopharm Tramadol HCl Once-A-Day (OAD) 200 mg film-coated tablets, and the reference product, Labopharm Tramadol HCl OAD 200 mg uncoated tablets, are bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects 18 to 55 years of age (inclusive).
* Body mass within 10% of the ideal mass in relation to height and age, according to the Body Mass Index (BMI).
* Body mass not less than 60 kg.
* Findings within the range of clinical acceptability in medical history and physical examination, and laboratory results within the "normal ranges" for the relevant laboratory tests (unless the investigator considered the deviation to be irrelevant for the purpose of the study).
* Normal electrocardiogram (ECG) and vital signs, or abnormalities which the investigator did not consider a disqualification for participation in the study.
* Willingness to undergo a pre-study physical examination and pre- and post-study laboratory investigations.
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and phase-related procedures).
* Non-smoker or past smoker who stopped smoking at least 3 months before entering the study.
* For females, the following conditions were to be met:

  * had been postmenopausal for at least 2 years, or
  * had been surgically sterilized, or
  * was of childbearing potential, and all of the following conditions were met:

    * had a normal menstrual flow within 1 month before study entry, and
    * had negative serum pregnancy test at screening. If this test was positive, the subject was to have been excluded from the study before receiving study medication. In the rare circumstance that a pregnancy was discovered after the subjects received study drug, then every attempt must be made to follow such subjects to term, and
    * must agree to use an accepted method of contraception (i.e., spermicide and barrier methods or spermicide and Intrauterine Device (IUD)). The subject had to agree to continue with the same method throughout the study. Hormonal contraceptives will not be allowed.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* History of, or current compulsive alcohol abuse (>10 drinks weekly), or regular exposure to other substances of abuse.
* Use of any medication, prescribed or over-the-counter, within 2 weeks prior to the first administration of study medication except if this would not have affected the outcome of the study in the opinion of the clinical investigator. Use of hormonal contraceptive agents by females were not allowed.
* Participation in another study with an experimental drug within 8 weeks before the first administration of study medication.
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system with evidence to this effect.
* A major illness during the 3 months before commencement of the screening period.
* History of hypersensitivity to the study drug or any related drugs.
* History of bronchial asthma.
* History of epilepsy.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of study medication.
* Diagnosis of hypotension made during the screening period.
* Diagnosis of hypertension made during the screening period or current diagnosis of hypertension.
* Resting pulse of >100 beats per minute or <45 beats per minute during the screening period, either supine or standing.
* Positive testing for hepatitis B antigen.
* Significant liver disease, defined as active hepatitis or elevated liver enzymes (e.g., AST (aspartate aminotransferase), Alanine transaminase (ALT)) >2 times the upper boundary of the normal range.
* Positive urine screen for drugs of abuse.
* Positive urine screen for tobacco use (SureStepTM Smoke Check Tests and One-Step Cotinine (COT) Tests).
* A serum pregnancy test (beta-hCG) either positive or not performed or lactation.
* History of marijuana, barbiturate, amphetamine or narcotic abuse within 12 months prior to study start.
* Participation in a tramadol study within the previous 12 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

REFERENCES:
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Started | 13 | 13
Completed | 12 | 12
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Treatment Period 2
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 13 | 13 | 26.0
  >=65 years | 0 | 0 | 0.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11.0
  Male | 7 | 8 | 15.0

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-t)
Description: Area under plasma concentration versus time curve to the last measurable concentration. Unit is ng.h/mL. h=hours.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Number analyzed (Participants) | 12 | 12
ng.h/mL | 5181 (1338) | 5010 (1176)

2. Secondary Outcome: Tmax
Description: Time to the maximum concentration
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Number analyzed (Participants) | 12 | 12
hours | 6 [3 to 12] | 6 [3 to 10]

3. Primary Outcome: AUC(0-Inf)
Description: Area under plasma concentration versus time curve extrapolated to infinity. Unit is ng.h/mL. h=hour.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Number analyzed (Participants) | 12 | 12
ng.h/mL | 5328 (1421) | 5175 (1241)

4. Primary Outcome: Cmax
Description: Maximum plasma concentration
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Number analyzed (Participants) | 12 | 12
ng/mL | 218 (49) | 209 (45)

5. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Number analyzed (Participants) | 12 | 12
hours | 7.08 (1.45) | 7.38 (1.76)

ADVERSE EVENTS:
Arm/Group | Tramadol HCl 200 mg Film-coated Tablets | Tramadol HCl 200 mg Uncoated Tablets
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 9/25 | 10/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol HCl 200 mg Film-coated Tablets (N=25) | Tramadol HCl 200 mg Uncoated Tablets (N=25)
Drowsiness (Nervous system disorders) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 7 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication based on the results of this study is envisaged, approval from the sponsor will be obtained and a draft manuscript will be submitted to the sponsor for scrutiny and comment.